CLINICAL TRIAL: NCT01888601
Title: TRAcking Non-small Cell Lung Cancer Evolution Through Therapy (Rx)
Acronym: TRACERx
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: UCL/12/0279
Record Dates: First submitted 2013-06-17; First posted 2013-06-28 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue, blood, plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NSCLC eligible for primary surgery: NSCLC eligible for primary surgery

SUMMARY:
To study the NSCLC evolutionary genomic landscape between primary and metastatic sites and the dynamics of intratumour heterogeneity over time combined with detailed clinical, histopathological and cancer phenotypic annotation for each patient, in order to significantly improve the outcomes of NSCLC patients (e.g. reduce their chance of recurrence and improve survival).

DETAILED DESCRIPTION:
The importance of intratumour genetic and functional heterogeneity is increasingly recognised as a driver of cancer progression and survival outcome. Understanding how tumour clonal heterogeneity impacts upon therapeutic outcome, however, is still an area of unmet clinical and scientific need. TRACERx (TRAcking non-small cell lung Cancer Evolution through therapy [Rx]), a prospective study of patients with primary non-small cell lung cancer (NSCLC), aims to define the evolutionary trajectories of lung cancer in both space and time through multiregion and longitudinal tumour sampling and genetic analysis. By following cancers from diagnosis to relapse, tracking the evolutionary trajectories of tumours in relation to therapeutic interventions, and determining the impact of clonal heterogeneity on clinical outcomes, TRACERx may help to identify novel therapeutic targets for NSCLC and may also serve as a model applicable to other cancer types.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent
* Patients ≥18 years of age, with early stage IIA-IIIB disease (according to TNM 8th edition) who are eligible for primary surgery. Patients with a radiological staging of IB (N0) who could be upstaged to IIA-IIIB following surgery (due to the presence of possible nodal involvement on the pre-operative scan) may also be included, but will be withdrawn if post-surgical staging remains IB.

Histopathologically confirmed NSCLC, or a strong suspicion of cancer on lung imaging necessitating surgery (e.g. diagnosis determined from frozen section in theatre)

* Primary surgery in keeping with NICE guidelines planned (see section 9.3)
* Agreement to be followed up at a TRACERx site
* Performance status 0 or 1
* Minimum tumour diameter at least 15mm to allow for sampling of at least two tumour regions (if 15mm, a high likelihood of nodal involvement on pre-operative imaging required to meet eligibility according to stage, i.e. T1N1-3)

Exclusion Criteria:

* Any other* malignancy diagnosed or relapsed at any time, which is currently being treated (including by hormonal therapy).
* Any other* current malignancy or malignancy diagnosed or relapsed within the past 3 years**.

  *Exceptions are: non-melanomatous skin cancer, stage 0 melanoma in situ, and in situ cervical cancer

  **An exception will be made for malignancies diagnosed or relapsed more than 2, but less than 3, years ago only if a pre-operative biopsy of the lung lesion has confirmed a diagnosis of NSCLC.
* Psychological condition that would preclude informed consent
* Treatment with neo-adjuvant therapy for current lung malignancy deemed necessary
* Post-surgery staging is not IIA-IIIB
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or syphilis infection.
* Sufficient tissue, i.e. a minimum of two tumour regions, is unlikely to be obtained for the study based on pre-operative imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage I-IIIA NSCLC eligible for primary surgery
Sampling Method: Non-Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2014-04; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intratumour heterogeneity | Year 5
  • Define the relationship between intratumour heterogeneity and clinical outcome following surgery and adjuvant therapy (including relationships between intratumour heterogeneity and clinical disease stage and histological subtypes of NSCLC).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Swanton, Principal Investigator — Chief Investigator
Locations (18):
- United Kingdom (18):
  - The Princess Alexandra Hospital NHS Trust, Harlow, Essex
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - University College London Hospitals NHS Foundation Trust, London, Select Region
  - Ashford and St Peter's Hospitals NHS Foundation Trust, Chertsey, Surrey
  - Grampian Health Board, Aberdeen
  - Heart of England NHS Foundation Trust, Birmingham
  - Cardiff and Vale University Health Board, Cardiff
  - NHS Greater Glasgow & Clyde, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Barts Health NHS Trust, London
  - North Middlesex University Hospital NHS Trust, London
  - The Whittington Hospital NHS Trust, trading as Whittington Health, London
  - Royal Free Hospital, London
  - Royal Free London NHS Foundation Trust - Barnet Hospital, London
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - University Hospital of South Manchester NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- [Derived] Biswas D, Liu YH, Herrero J, Wu Y, Moore DA, Karasaki T, Grigoriadis K, Lu WT, Veeriah S, Naceur-Lombardelli C, Magno N, Ward S, Frankell AM, Hill MS, Colliver E, de Carne Trecesson S, East P, Malhi A, Snell DM, O'Neill O, Leonce D, Mattsson J, Lindberg A, Micke P, Moldvay J, Megyesfalvi Z, Dome B, Fillinger J, Nicod J, Downward J, Szallasi Z; TRACERx Consortium; Hackshaw A, Jamal-Hanjani M, Kanu N, Birkbak NJ, Swanton C. Prospective validation of ORACLE, a clonal expression biomarker associated with survival of patients with lung adenocarcinoma. Nat Cancer. 2025 Jan;6(1):86-101. doi: 10.1038/s43018-024-00883-1. Epub 2025 Jan 9. PMID 39789179
- [Derived] Pan X, AbdulJabbar K, Coelho-Lima J, Grapa AI, Zhang H, Cheung AHK, Baena J, Karasaki T, Wilson CR, Sereno M, Veeriah S, Aitken SJ, Hackshaw A, Nicholson AG, Jamal-Hanjani M; TRACERx Consortium; Swanton C, Yuan Y, Le Quesne J, Moore DA. The artificial intelligence-based model ANORAK improves histopathological grading of lung adenocarcinoma. Nat Cancer. 2024 Feb;5(2):347-363. doi: 10.1038/s43018-023-00694-w. Epub 2024 Jan 10. PMID 38200244
- [Derived] Abbosh C, Frankell AM, Harrison T, Kisistok J, Garnett A, Johnson L, Veeriah S, Moreau M, Chesh A, Chaunzwa TL, Weiss J, Schroeder MR, Ward S, Grigoriadis K, Shahpurwalla A, Litchfield K, Puttick C, Biswas D, Karasaki T, Black JRM, Martinez-Ruiz C, Bakir MA, Pich O, Watkins TBK, Lim EL, Huebner A, Moore DA, Godin-Heymann N, L'Hernault A, Bye H, Odell A, Kalavakur P, Gomes F, Patel AJ, Manzano E, Hiley CT, Carey N, Riley J, Cook DE, Hodgson D, Stetson D, Barrett JC, Kortlever RM, Evan GI, Hackshaw A, Daber RD, Shaw JA, Aerts HJWL, Licon A, Stahl J, Jamal-Hanjani M; TRACERx Consortium; Birkbak NJ, McGranahan N, Swanton C. Tracking early lung cancer metastatic dissemination in TRACERx using ctDNA. Nature. 2023 Apr;616(7957):553-562. doi: 10.1038/s41586-023-05776-4. Epub 2023 Apr 13. PMID 37055640
- [Derived] Frankell AM, Dietzen M, Al Bakir M, Lim EL, Karasaki T, Ward S, Veeriah S, Colliver E, Huebner A, Bunkum A, Hill MS, Grigoriadis K, Moore DA, Black JRM, Liu WK, Thol K, Pich O, Watkins TBK, Naceur-Lombardelli C, Cook DE, Salgado R, Wilson GA, Bailey C, Angelova M, Bentham R, Martinez-Ruiz C, Abbosh C, Nicholson AG, Le Quesne J, Biswas D, Rosenthal R, Puttick C, Hessey S, Lee C, Prymas P, Toncheva A, Smith J, Xing W, Nicod J, Price G, Kerr KM, Naidu B, Middleton G, Blyth KG, Fennell DA, Forster MD, Lee SM, Falzon M, Hewish M, Shackcloth MJ, Lim E, Benafif S, Russell P, Boleti E, Krebs MG, Lester JF, Papadatos-Pastos D, Ahmad T, Thakrar RM, Lawrence D, Navani N, Janes SM, Dive C, Blackhall FH, Summers Y, Cave J, Marafioti T, Herrero J, Quezada SA, Peggs KS, Schwarz RF, Van Loo P, Miedema DM, Birkbak NJ, Hiley CT, Hackshaw A, Zaccaria S; TRACERx Consortium; Jamal-Hanjani M, McGranahan N, Swanton C. The evolution of lung cancer and impact of subclonal selection in TRACERx. Nature. 2023 Apr;616(7957):525-533. doi: 10.1038/s41586-023-05783-5. Epub 2023 Apr 12. PMID 37046096
- [Derived] Al Bakir M, Huebner A, Martinez-Ruiz C, Grigoriadis K, Watkins TBK, Pich O, Moore DA, Veeriah S, Ward S, Laycock J, Johnson D, Rowan A, Razaq M, Akther M, Naceur-Lombardelli C, Prymas P, Toncheva A, Hessey S, Dietzen M, Colliver E, Frankell AM, Bunkum A, Lim EL, Karasaki T, Abbosh C, Hiley CT, Hill MS, Cook DE, Wilson GA, Salgado R, Nye E, Stone RK, Fennell DA, Price G, Kerr KM, Naidu B, Middleton G, Summers Y, Lindsay CR, Blackhall FH, Cave J, Blyth KG, Nair A, Ahmed A, Taylor MN, Procter AJ, Falzon M, Lawrence D, Navani N, Thakrar RM, Janes SM, Papadatos-Pastos D, Forster MD, Lee SM, Ahmad T, Quezada SA, Peggs KS, Van Loo P, Dive C, Hackshaw A, Birkbak NJ, Zaccaria S; TRACERx Consortium; Jamal-Hanjani M, McGranahan N, Swanton C. The evolution of non-small cell lung cancer metastases in TRACERx. Nature. 2023 Apr;616(7957):534-542. doi: 10.1038/s41586-023-05729-x. Epub 2023 Apr 12. PMID 37046095
- [Derived] Ng KW, Boumelha J, Enfield KSS, Almagro J, Cha H, Pich O, Karasaki T, Moore DA, Salgado R, Sivakumar M, Young G, Molina-Arcas M, de Carne Trecesson S, Anastasiou P, Fendler A, Au L, Shepherd STC, Martinez-Ruiz C, Puttick C, Black JRM, Watkins TBK, Kim H, Shim S, Faulkner N, Attig J, Veeriah S, Magno N, Ward S, Frankell AM, Al Bakir M, Lim EL, Hill MS, Wilson GA, Cook DE, Birkbak NJ, Behrens A, Yousaf N, Popat S, Hackshaw A; TRACERx Consortium; CAPTURE Consortium; Hiley CT, Litchfield K, McGranahan N, Jamal-Hanjani M, Larkin J, Lee SH, Turajlic S, Swanton C, Downward J, Kassiotis G. Antibodies against endogenous retroviruses promote lung cancer immunotherapy. Nature. 2023 Apr;616(7957):563-573. doi: 10.1038/s41586-023-05771-9. Epub 2023 Apr 12. PMID 37046094
- [Derived] Martinez-Ruiz C, Black JRM, Puttick C, Hill MS, Demeulemeester J, Larose Cadieux E, Thol K, Jones TP, Veeriah S, Naceur-Lombardelli C, Toncheva A, Prymas P, Rowan A, Ward S, Cubitt L, Athanasopoulou F, Pich O, Karasaki T, Moore DA, Salgado R, Colliver E, Castignani C, Dietzen M, Huebner A, Al Bakir M, Tanic M, Watkins TBK, Lim EL, Al-Rashed AM, Lang D, Clements J, Cook DE, Rosenthal R, Wilson GA, Frankell AM, de Carne Trecesson S, East P, Kanu N, Litchfield K, Birkbak NJ, Hackshaw A, Beck S, Van Loo P, Jamal-Hanjani M; TRACERx Consortium; Swanton C, McGranahan N. Genomic-transcriptomic evolution in lung cancer and metastasis. Nature. 2023 Apr;616(7957):543-552. doi: 10.1038/s41586-023-05706-4. Epub 2023 Apr 12. PMID 37046093
- [Derived] AbdulJabbar K, Raza SEA, Rosenthal R, Jamal-Hanjani M, Veeriah S, Akarca A, Lund T, Moore DA, Salgado R, Al Bakir M, Zapata L, Hiley CT, Officer L, Sereno M, Smith CR, Loi S, Hackshaw A, Marafioti T, Quezada SA, McGranahan N, Le Quesne J; TRACERx Consortium; Swanton C, Yuan Y. Geospatial immune variability illuminates differential evolution of lung adenocarcinoma. Nat Med. 2020 Jul;26(7):1054-1062. doi: 10.1038/s41591-020-0900-x. Epub 2020 May 27. PMID 32461698
- [Derived] Hynds RE, Ben Aissa A, Gowers KHC, Watkins TBK, Bosshard-Carter L, Rowan AJ, Veeriah S, Wilson GA, Quezada SA, Swanton C; TRACERx Consortium; Janes SM. Expansion of airway basal epithelial cells from primary human non-small cell lung cancer tumors. Int J Cancer. 2018 Jul 1;143(1):160-166. doi: 10.1002/ijc.31383. Epub 2018 Apr 6. PMID 29569246
- [Derived] Jamal-Hanjani M, Wilson GA, McGranahan N, Birkbak NJ, Watkins TBK, Veeriah S, Shafi S, Johnson DH, Mitter R, Rosenthal R, Salm M, Horswell S, Escudero M, Matthews N, Rowan A, Chambers T, Moore DA, Turajlic S, Xu H, Lee SM, Forster MD, Ahmad T, Hiley CT, Abbosh C, Falzon M, Borg E, Marafioti T, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Shah R, Joseph L, Quinn AM, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Dentro S, Taniere P, O'Sullivan B, Lowe HL, Hartley JA, Iles N, Bell H, Ngai Y, Shaw JA, Herrero J, Szallasi Z, Schwarz RF, Stewart A, Quezada SA, Le Quesne J, Van Loo P, Dive C, Hackshaw A, Swanton C; TRACERx Consortium. Tracking the Evolution of Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Jun 1;376(22):2109-2121. doi: 10.1056/NEJMoa1616288. Epub 2017 Apr 26. PMID 28445112